CLINICAL TRIAL: NCT01570790
Title: An Open Label, Pilot (Phase I/II), Dose-Escalation Safety and Tolerability Study of Combretastatin A4 Phosphate in Patients With Neovascular Age-Related Macular Degeneration.
Brief Title: Combretastatin A4 Phosphate in Patients With Neovascular Age-Related Macular Degeneration
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FBO-206
Record Dates: First submitted 2012-04-02; First posted 2012-04-04 (Estimated); Last update posted 2017-12-06 (Actual); Status verified 2017-12

CONDITIONS: Combretastatin A4 Phosphate; Age-related Macular Degeneration; AMD; CNV; Choroidal Neovascularization
MeSH Terms: conditions — Macular Degeneration; Choroidal Neovascularization | interventions — fosbretabulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort 1 (Experimental)
  Interventions: Drug: Combretastatin A-4 phosphate
- Cohort 2 (Experimental)
  Interventions: Drug: Combretastatin A-4 Phosphate
- Cohort 3 (Experimental)
  Interventions: Drug: Combretastatin A-4 Phosphate

INTERVENTIONS:
Drug: Combretastatin A-4 phosphate — 27 mg/m2 CA4P IV infusion at baseline and every week for 4 doses
  Other Names: fosbretabulin disodium
  Arms: Cohort 1
Drug: Combretastatin A-4 Phosphate — 36 mg/m2 CA4P IV infusion at baseline and every week for 4 doses
  Other Names: fosbretabulin disodium
  Arms: Cohort 2
Drug: Combretastatin A-4 Phosphate — 45 mg/m2 CA4P IV infusion at baseline and every week for 4 doses
  Other Names: fosbretabulin disodium
  Arms: Cohort 3

SUMMARY:
The purpose of the study is assess safety, bioactivity, and maximal tolerated dose of repeated weekly intravenous infusion of combretastatin A-4 phosphate (CA4P) in patients with neovascular age-related macular degeneration

DETAILED DESCRIPTION:
The study is designed as a single escalating dose with cohorts of five subjects. Escalation to the next cohort was based on the presence of no more than one subject with a dose limiting toxicity (DLT). The first cohort is to receive 27 mg/m2 intravenous infusion of of CA4P, 36mg/m2 to the second cohort, and 45mg/m2 to the third cohort. CA4P will be infused at baseline and every week for a total of 4 doses. Follow up visits will be scheduled at week 8 and 12.

Safety data will be collected during the 12-week duration of the study and will be assessed using the common terminology criteria of adverse events (CTCAE v3.0). Bioactivity data will be assessed by measuring change in best corrected visual acuity, changes in central retinal thickness as measured by Optical coherence tomography, and changes in the amount of leakage on fluorescein angiography.

DLTs were defined as specific events that are considered to be probably or definitely related to CA4P. Major DLTs included QTc interval ≥ 500 msec (based on measurements provided by the core laboratory for ECG analysis), Grade-2 or greater ventricular arrhythmia, unexplained syncope, Grade-3 or greater toxicity, delayed recovery postponing re-treatment by >14 days, and ocular toxicity such as keratopathy, uveitis, optic neuropathy, and retinopathy, at the discretion of the investigator.

ELIGIBILITY:
Inclusion Criteria:

1. Age 50 years or older;
2. 12-lead electrocardiogram (ECG) performed at least 2 weeks but less than 4 weeks prior to entry into the study showing a QTc <440 with no evidence of current or prior myocardial ischemia, infarction or significant arrhythmia as determined by review and signature of the cardiologist.
3. Adequate bone marrow function:

   Absolute granulocyte count ≥1500 cells/mm3; Platelet count ≥100,000 cells/mm3; Hemoglobin ≥9.0gm/ dL;
4. PT/PTT within the institution upper limit of normal (ULN) or INR <1.1 ;
5. Adequate hepatic function:

   Total bilirubin within the institution ULN; Alanine and aspartate aminotransferase (ALT/AST) <3 times the institutional ULN;
6. Adequate renal function: serum creatinine ≤2.0 mg/dL;
7. Ophthalmic criteria:

   1. Best corrected visual acuity in the study eye of ≤20/40 and ≥20/800 in the fellow eye.
   2. Subfoveal choroidal neovascularization (as illustrated by fluorescein angiography) secondary to age-related macular degeneration, with a total lesion size of ≤12 total disc areas, of which at least 50% must be active CNV.
   3. Subretinal hemorrhage ≤50% of total lesion size;
   4. For patients with minimally classic and purely occult CNV, there must be documented evidence of ≥2 lines of vision loss (ETDRS) during the previous 12 weeks;
   5. Clear ocular media and adequate papillary dilatation to permit good quality stereoscopic fundus photography;
8. Male fertile patients must abstain from sexual intercourse or use effective birth control;
9. Women must be post-menopausal for at least 12 months prior to study entry, or surgically sterile, or must be using two forms of effective contraception.
10. Able to return for all study visits within required visit windows;
11. Be able to give written informed consent.

Exclusion Criteria:

1. Previous subfoveal thermal laser therapy;
2. Any subfoveal scarring or atrophy, or >25% of the total lesion size is made up of scarring or atrophy;
3. Significant media opacities, including cataract, which can interfere with visual acuity, assessment of toxicity, or fundus photography;
4. Presence of other causes of choroidal neovascularization, including pathologic myopia (spherical equivalent of ≥-8.0 diopters, or axial length of ≥25mm), ocular histoplasmosis syndrome, angioid streaks, choroidal rupture, and multifocal choroiditis and other uveitic entities;
5. Any condition that might interfere with assessment of the progression of CNV;
6. Any intraocular surgery in the study eye within 12 weeks of screening for the study;
7. Other treatment for AMD of the study eye within 12 weeks prior to screening;
8. Known allergy to fluorescein;
9. Any current or history of significant gastrointestinal, oral, or nasal bleeding;
10. Serious intercurrent infections or other nonmalignant medical illnesses that are uncontrolled or whose control may be jeopardized by the complications of this therapy;
11. Grade 2 (CTC v.3.0) or greater pre-existing peripheral neuropathy;
12. Psychiatric disorders or other conditions rendering patients incapable of complying with the requirements of the protocol;
13. Pregnant or breast-feeding women;
14. History of angina, myocardial infarction, CHF, non-controlled atrial arrhythmias or clinically significant arrhythmias including conduction abnormality, nodal junctional arrhythmias and dysrhythmias, sinus bradycardia or tachycardia, supraventricular arrhythmias, atrial fibrillation or flutter, syncope or vasovagal episodes;
15. Abnormal cardiac stress test;
16. Uncontrolled hypertension (consistently >150/100mmHg irrespective of medication);
17. Uncontrolled hypokalemia and/or hypomagnesemia;
18. ECG with evidence of prior myocardial infarction, QTc > 450 msec or other clinically significant abnormalities;
19. Drug(s) known to prolong the QTc interval;
20. Patients with conditions associated with QTc prolongation;
21. Any investigational drug or device within 4 weeks prior to screening;
22. Decreased ejection fraction ≤50% or prior myocardial infarction.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2003-05; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability | 12 weeks after the first infusion of the Study Drug
  To report frequency and severity of adverse events, as defined by the common terminology criteria of adverse events (CTCAE v.3.0; National Cancer Institute), and to determine the degree of relationship of adverse events to the study drug (CA4P).
Dose Limiting Toxicities (DLT) | 12 weeks after the first infusion of the study drug
  DLT is defined as any of the following adverse events if ≥Grade-2 in severity: ventricular arrhythmia, second or third degree AV block, severe sinus bradycardia < 45 bpm, tachycardia >120 bpm, supraventricular arrhythmia > 24 hours, ventricular tachycardia (>9 beats in a row), any length of torsades de pointes, unexplained recurrent syncope, QTc prolongation ≥500 msec on > 2 consecutive ECGs, Grade-2 or greater myocardial infarction, or ocular toxicities deemed by the investigator not acceptable for the patients to receive further treatments.

SECONDARY OUTCOMES:
Maximum Tolerated Dose | 12 weeks after the first infusion of the study drug
  Maximum Tolerated Dose (MTD) of intravenous infusion of combretastatin A-4 phosphate in patients with neovascular age related macular degeneration. The MTD is defined as the maximum dose level of CA4P administered at which, DLT is observed in fewer than 2 patients at a given cohort.
Change in Best Corrected Visual Acuity | 4 and 12 weeks after first infusion of the study drug
  Difference change from baseline in Best corrected visual acuity, as measured using the Early Treatment Diabetic Retinopathy Study (ETDRS) protocol, at week 4 and week 12.
Change in Central Retinal Thickness | 4 and 12 weeks following the first infusion of CA4P
  Difference change from baseline in central retinal thickness as measured by Optical Coherence Tomography at week 4 and week 12.

CONTACTS AND LOCATIONS:
Overall Officials: Quan D Nguyen, MD, MSc, Principal Investigator — Wilmer Eye Institute - Johns Hopkins University School of Medicine
Locations (1):
- Wilmer Eye Institute, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Ibrahim MA, Do DV, Sepah YJ, Shah SM, Van Anden E, Hafiz G, Donahue JK, Rivers R, Balkissoon J, Handa JT, Campochiaro PA, Nguyen QD. Vascular disrupting agent for neovascular age related macular degeneration: a pilot study of the safety and efficacy of intravenous combretastatin A-4 phosphate. BMC Pharmacol Toxicol. 2013 Jan 14;14:7. doi: 10.1186/2050-6511-14-7. PMID 23316779